CLINICAL TRIAL: NCT04705077
Title: A Phase 1, Open-Label Study to Assess the Single Dose Pharmacokinetics of Suspension and Capsule Formulations of SR419 and Repeat Dose Pharmacokinetics of Capsule Formulation of SR419, and to Assess the Effect of a High-Fat Meal on the Pharmacokinetics of SR419 in Healthy Subjects
Brief Title: A Study to Assess the Pharmacokinetics and Food Effect of SR419 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SIMR (Australia) Biotech Pty Ltd. (Industry)
Responsible Party: Sponsor
Organization: SIMRAustraliaBiotech (Unknown)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SR419-103
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Dose Treatment (Experimental): Each subject will be assigned to the fixed period sequence.
  * Period 1: SR419 suspension in the fasted state;
  * Period 2: SR419 capsule in the fasted state;
  * Period 3: SR419 capsule in the fed state (high-fat meal).
  Interventions: Drug: SR419
- Repeated Dose Treatment (Experimental): Each subject will receive 30 mg of SR419 capsule, once every 8 hours (Q8h), for 5 days.
  Interventions: Drug: SR419

INTERVENTIONS:
Drug: SR419 — 2 formulations of SR419, SR419 suspension and SR419 capsule will be used in the study.

SUMMARY:
This will be an open-label, single-site, Phase I study to evaluate the PK, safety, and tolerability of SR419 in healthy volunteers.

DETAILED DESCRIPTION:
This study is a phase 1, open-label study to assess the single dose pharmacokinetics of suspension and capsule formulations of SR419 and repeat dose pharmacokinetics of capsule formulation of SR419, and to assess the effect of a high-fat meal on the pharmacokinetics of SR419 in healthy subjects.The trial will consist of 3 cohorts. Cohort 1 and 2 will follow a single sequence, 3-period, 2-formulation, dosing in fasted or fed state design. Cohort 3 will be a repeated dose study of SR419 capsule in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females who are 18 to 64 years of age inclusive, are eligible.
2. Body weight > 50 kg (110 pounds) and body mass index (BMI) between 18 and 30 kg/m2.
3. Male or female subjects must agree to use contraception methods.
4. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

1. Clinically significant history of central nervous system (CNS) disease.
2. Current or chronic history of liver disease or known hepatic or biliary abnormalities
3. History of regular alcohol consumption within 6 months of screening defined as: an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~285 mL) of beer, 1 glass (125 mL) of wine or 1 measure (25 mL) of spirits.
4. History of significant drug abuse within one year of screening or use of soft drugs (such as marijuana) within 3 months prior to screening or hard drugs (such as cocaine, methamphetamine, crack) within 1 year prior to screening.
5. History of sensitivity to any of the components thereof or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates participation.
6. History of asthma (excluding resolved childhood asthma), anaphylaxis or anaphylactoid reactions, severe allergic responses.
7. History of hypercoagulable state or history of thrombosis.
8. A positive Hepatitis B surface antigen, Hepatitis C antibody or human immunodeficiency virus (HIV) antibody result.
9. A positive urinary cotinine test or history of regular use of tobacco- or nicotine-containing products (more than 4 products per month within 6 months prior to screening) or unwilling to refrain from use of such products from Screening until completion of the final study visit.
10. A positive drug/alcohol result.
11. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
12. Unable to refrain from consumption of Seville oranges, grapefruit or grapefruit juice within 7 days prior to the first dose of IMP until the Safety Follow-up visit.
13. A positive pregnancy test result.
14. Breast-feeding and/or lactating subject.
15. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration of SR419 | Up to Day 12
Time of peak plasma concentration of SR419 | Up to Day 12
Area under the plasma concentration-time curve of SR419 | Up to Day 12
Apparent total clearance of SR419 | Up to Day 12
Terminal half-life of SR419 | Up to Day 12
Accumulation ratio of SR419 | Up to Day 12

SECONDARY OUTCOMES:
Peak plasma concentration of SR419 metabolites | Up to Day 12
Time of peak plasma concentration of SR419 metabolites | Up to Day 12
Area under the plasma concentration-time curve of SR419 metabolites | Up to Day 12
Terminal half-life of SR419 metabolites | Up to Day 12
Accumulation ratio of SR419 metabolites | Up to Day 12
Number of participants with adverse events | Up to Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Polasek, Principal Investigator — CMAX Clinical Research
Locations (1):
- CMAX Clinical Research, Adelaide, Australia

IPD SHARING:
Plan to Share IPD: No